CLINICAL TRIAL: NCT04393636
Title: Randomized Controlled Trial of Digital Cardiac Counseling in Patients With Delayed Cardiac Surgical Treatment Due to Covid-19 Pandemic (DCC Trial)
Brief Title: Digital Cardiac Counseling Trial: DCC Trial
Acronym: DCC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Ziekenhuis Maastricht (Other)
Responsible Party: Principal Investigator, Peyman Sardari Nia, Principal investigator, Academisch Ziekenhuis Maastricht
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NL72754.068.20
Record Dates: First submitted 2020-05-11; First posted 2020-05-19 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Cardiovascular Diseases; Cardiovascular Risk Factor
Keywords: Digital Cardiac Counseling; Prehabilitation; cardiac surgical waiting list
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Preoperative Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control arm (No Intervention): Participants will receive at the different time intervals through our custom-made Digital Cardiac Counselling platform different questionnaires related to the different known risk factors for the perioperative cardiac care and measured outcomes.Additional to known risk factors a Covid-19 module will be used as well.
- Intervention arm (Active Comparator): All participants will receive at the different time intervals through our custom-made Digital Cardiac Counseling platform different questionnaires related to the different known risk factors for the perioperative cardiac care and measured outcomes. Additional to above participants in the intervention group will receive through the Digital Cardiac Counseling platform different modules with E-counseling for risk factors evaluated in the questionnaires. Additional to known risk factors a Covid-19 module will be used as well.
  Interventions: Other: Digital cardiac Counseling

INTERVENTIONS:
Other: Digital cardiac Counseling — * Screening for reduced physical fitness and digital counseling.
  * Screening for smoking and digital counseling.
  * Screening for malnutrition and obesity and digital counseling.
  * Screening for anxiety and depression and digital counseling.
  * Screening for elevated pulmonary risk score and digital counseling.
  Other Names: prehabilitation
  Arms: Intervention arm

SUMMARY:
Most patients undergoing a cardiovascular procedure need an ICU-bed during the hospitalization and therefore it is possible that for the unforeseen future, because of the Covid-19 crisis, many patients will stay on the waiting list for many months to come. There are some studies showing an increased mortality associated with an increased waiting time for the patients on the waiting list for an elective cardiac surgery. However, there is no data on the evolution of the morbidity, the quality of life and the symptomatology of the patients waiting for an elective operation. Also it is not clear whether the period of waiting for an elective cardiovascular operation would impact the morbidity or the mortality of the planned operation at later stage. Furthermore, there is a plethora of studies on risk factors associated with the perioperative morbidity and mortality in general. Therefore, the rationale of the current study is to evaluate whether Digital Cardiac Counseling (DCC) would improve outcomes of the patients waiting for an elective cardiac operation. At the DCC platform, there will be assessments of cardiovascular symptoms, Covid-19 prevention for cardiovascular patients, smoking cessation, anxiety relief, exercise stimulation, pulmonary rehabilitation and diet adjustments. This will be done by means of questionnaires and E-consults.

DETAILED DESCRIPTION:
Rationale:

Most patients undergoing a cardiovascular procedure need an ICU-bed during the hospitalization and therefore it is possible that for the unforeseen future, because of the Covid-19 crisis, many patients will stay on the waiting list for many months to come. There are some studies showing an increased mortality associated with an increased waiting time for the patients on the waiting list for an elective cardiac surgery. However, there is no data on the evolution of the morbidity, the quality of life and the symptomatology of the patients waiting for an elective operation. Also it is not clear whether the period of waiting for an elective cardiovascular operation would impact the morbidity or the mortality of the planned operation at later stage. Furthermore, there is a plethora of studies on risk factors associated with the perioperative morbidity and mortality in general. Therefore, the rationale of the current study is to evaluate whether Digital Cardiac Counseling (DCC) would improve outcomes of the patients waiting for an elective cardiac operation. At the DCC platform, there will be assessments of cardiovascular symptoms, Covid-19 prevention for cardiovascular patients, smoking cessation, anxiety relief, exercise stimulation, pulmonary rehabilitation and diet adjustments. This will be done by means of questionnaires and E-consults. Investigators start this project now because of two reasons. First, the prolonged waiting list due to the Covid pandemic creates the opportunity to use this period for cardiac prehabilitation. Second, it is only recently that the investigators got the possibility to use a digital platform, which is ideal in this period of social distancing.

Objective:

Primary Objective:

* What is the effect of an interactive Digital Cardiac Counseling platform with E-consulting on cumulative incidence of major adverse cardiovascular events (MACE) at 1 year after the cardiac surgery compared to the control condition (no interactive Digital Cardiac Counseling)?

Secondary Objective(s): - What is the effect of an interactive Digital Cardiac Counseling platform with E-consulting on patient-measured outcomes during treatment delay due to the Covid-19 pandemic measured just before, and 1 year after the cardiac surgery compared to the control condition (no interactive Digital Cardiac Counseling)?

Study design:

Randomized controlled trial. The investigators will use random permuted block size if technically feasible otherwise with random block sizes of 4, 6, and 8. The randomization will be computer-based and will generate two groups. Both groups will get access to the Digital Cardiac Counseling platform and both groups will complete the same set of validated questionnaires at the same time intervals. The intervention groups will get additional training modules and E-consulting based on the risk assessment retrieved from the completed questionnaires.

Study population:

The patient population will include any adult patient on the waiting list for any elective cardiovascular operation in MUMC (Maastricht University Medical Center) during Covid-19 pandemic.

Intervention:

the intervention group will receive through the Digital Cardiac Counselling platform different modules with E-counselling for risk factors evaluated in the questionnaires.The digital counselling modules for intervention group are described below: -

* Screening for reduced physical fitness. If there are signs for a decreased physical condition we will refer the patient, after consultation, for a digital intake with our physiotherapist. The patients then get access to a digital module with information and videos of physical exercise training. The patient gets a trainings schedule and the investigators will contact the patient after about 1 and 3 weeks to check their progression and to give additional advice when needed.
* Screening for smoking. If the patient smokes and is motivated to quit smoking, the investigators will refer, after consultation, for a digital intake with one of our stop smoking nurses. Then, a digital and telephone supported counselling will start after an informed and shared decision making with the nurse. When needed, supportive medication can be prescribed.
* Screening for malnutrition and obesity. If there are signs of malnutrition (MUST-score) or obesity (BMI >30) the investigators will refer the patient, after consultation, for a digital intake with a dietician. The patients then get access to a digital module with information about a healthy diet. The investigators will contact the patient ever 2 weeks in case of malnutrition and every 4 weeks in case of obesity. In the case of malnutrition the dietician can prescribe protein rich nutrition supplements when needed.
* Screening for anxiety and depression. If there are signs for anxiety and depression, the investigators will refer the patient, after consultation, for a digital intake with a psychological assistant. The patients then get access to a digital platform with information and exercises. The psychological assistant will guide the patient and will provide digital support after 1 and 3 weeks.
* Screening for elevated pulmonary risk score. When patients have an elevated risk score for adverse pulmonary complications (pulmonary risk score for cardiac surgery patients questionnaire) the investigators will refer the patient, after consultation, for a digital intake with our physiotherapist. The patients then get access to a digital module with information and videos of pulmonary exercise training. The investigators will send a inspiratory muscle trainer (IMT) to the patient to perform daily exercises. The patient gets a trainings schedule and the investigators will contact the patient after about 1 and 3 weeks to check their progression and to give additional advice when needed.

Main study parameters/endpoints:

The primary endpoint is cumulative incidence of MACE (Major Adverse Cardiovascular Events) at 1 year after cardiac surgery. The primary outcome is the difference in percentage of patients that experienced Mace at 1-year follow-up postoperatively. The investigators expect that approximately 20% of patients in the control group will experience an event. The investigators will include 197 patients per group, or 394 in total, to be able to have 80% power to detect a difference in MACE of 10% between groups in favor of the intervention group, using an alpha of 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are on the waiting list for any elective cardiac operation and are older than 18 years old (adult cardiac surgery patients) during the Covid-19 pandemic
* Patients accepted for any elective cardiac operation and are older than 18 years during the Covid-19 pandemic (adult cardiac surgery patients)

Exclusion Criteria:

* Patients who are not able to use digital platforms for various reasons (blindness, illiteracy, neurological deficits, mental inability etc.)
* Patients who do not have an Internet connection or any digital platform and whose direct family are not able to provide that.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 394 (Actual)
Dates: Start 2020-06-05 (Actual); Primary Completion 2024-03-22 (Actual); Study Completion 2024-03-22 (Actual)

PRIMARY OUTCOMES:
MACEs | Cumulative incidence (from inclusion) at 1 year postoperatively
  Major Adverse Cardiovascular Events defined as Cardiovascular death, non-fatal myocardial infarction, non-fatal stroke, hospitalization for heart failure and/or fo earlier planned intervention

SECONDARY OUTCOMES:
Mortality | Before the scheduled date of the operation, at 30 days, in-hospital (at 30 days or during the same hospitalization for the planned procedure), at one-year postoperatively and cumulative from inclusion at 1-year postoperatively
  all-cause mortality
Cardiovascular-related mortality | Before the scheduled date of the operation, at one-year postoperatively and cumulative from inclusion at 1-year postoperatively
  Mortality caused by cardiovascular disease
Covid-19 related mortality | Before the scheduled date of the operation, at one-year postoperatively and cumulative from inclusion at 1-year postoperatively
  Mortality caused by Covid-19 infection and/or related complications
Health-related quality of life | during waiting time measured before the procedure, at 3 months, at 6 months and at 12 months
  Measured using SF (Short Form) 36 Health Survey
NYHA Functional classification | during waiting time measured before the procedure, at 3 months, at 6 months and at 12 months
  New York Heart Association Functional Classification
CCS (Canadian Cardiovascular Society grading of angina pectoris) | during waiting time measured before the procedure, at 3 months, at 6 months and at 12 months
  Grading of angina pectoris
MACEs | during waiting time measured before the scheduled date of the operation, at 1-year postoperatively
  Major Adverse Cardiovascular Events defined as Cardiovascular death, non-fatal myocardial infarction, non-fatal stroke, hospitalization for heart failure and/or fo earlier planned intervention
Perioperative complications | during waiting time measured before the scheduled date of the operation, at 30 days postoperatively and at 90 days postoperatively
  Respiratory failure, pneumonia, septicemia, renal failure, myocardial infarction, stroke, atrial fibrillation, pacemaker implantation, re-operation, delirium, wound infection, urinary tract infection and pressure ulcers
Hospital length of stay | from the admission to the hospital untill discharge from the hospital, assessed up to 12 months
  from surgery until discharge in days
Time on mechanical ventilation | from the admission to the ICU untill discharge from the ICU, assessed up to 12 months
  measured in hours from arrival in ICU until extubation
Smoking status | during waiting time measured before the procedure, at 3 months, at 6 months and at 12 months
  whether patient is active smoking
Anxiety and Depression | during waiting time measured before the procedure, at 3 months, at 6 months and at 12 months
  Measured using HADS (Hospital Anxiety and Depression Scale) score
Participation in postoperative cardiac rehabilitation | postoperatively at 3 months, at 6 months and at 12 months
  the percentage of patients taking part in postoperative cardiac rehabilitation
Body-Mass Index (BMI) | during waiting time measured before the procedure, at 3 months, at 6 months and at 12 months
  Percentage BMI<20 or BMI>30
Number of participants with unplanned visits | during waiting time measured before the procedure, at 3 months, at 6 months and at 12 months
  Unplanned visits to emergency department
Healthcare costs | during waiting time measured before the procedure, at 3 months, at 6 months and at 12 months
  Total costs of the whole treatment process

CONTACTS AND LOCATIONS:
Locations (1):
- Maastricht University Medical Center, Maastricht, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zheng YY, Ma YT, Zhang JY, Xie X. COVID-19 and the cardiovascular system. Nat Rev Cardiol. 2020 May;17(5):259-260. doi: 10.1038/s41569-020-0360-5. PMID 32139904
- [Result] Plomp J, Redekop WK, Dekker FW, van Geldorp TR, Haalebos MM, Jambroes G, Kingma JH, Zijlstra F, Tijssen JG. Death on the waiting list for cardiac surgery in The Netherlands in 1994 and 1995. Heart. 1999 Jun;81(6):593-7. doi: 10.1136/hrt.81.6.593. PMID 10336916
- [Result] Morgan CD, Sykora K, Naylor CD. Analysis of deaths while waiting for cardiac surgery among 29,293 consecutive patients in Ontario, Canada. The Steering Committee of the Cardiac Care Network of Ontario. Heart. 1998 Apr;79(4):345-9. PMID 9616340
- [Result] Malaisrie SC, McDonald E, Kruse J, Li Z, McGee EC Jr, Abicht TO, Russell H, McCarthy PM, Andrei AC. Mortality while waiting for aortic valve replacement. Ann Thorac Surg. 2014 Nov;98(5):1564-70; discussion 1570-1. doi: 10.1016/j.athoracsur.2014.06.040. Epub 2014 Sep 18. PMID 25240781
- [Result] da Fonseca VBP, De Lorenzo A, Tura BR, Pittella FJM, da Rocha ASC. Mortality and morbidity of patients on the waiting list for coronary artery bypass graft surgery. Interact Cardiovasc Thorac Surg. 2018 Jan 1;26(1):34-40. doi: 10.1093/icvts/ivx276. PMID 29049704
- [Result] Turner AJ, Hiscox JA, Hooper NM. ACE2: from vasopeptidase to SARS virus receptor. Trends Pharmacol Sci. 2004 Jun;25(6):291-4. doi: 10.1016/j.tips.2004.04.001. PMID 15165741
- [Result] Chan JF, Yuan S, Kok KH, To KK, Chu H, Yang J, Xing F, Liu J, Yip CC, Poon RW, Tsoi HW, Lo SK, Chan KH, Poon VK, Chan WM, Ip JD, Cai JP, Cheng VC, Chen H, Hui CK, Yuen KY. A familial cluster of pneumonia associated with the 2019 novel coronavirus indicating person-to-person transmission: a study of a family cluster. Lancet. 2020 Feb 15;395(10223):514-523. doi: 10.1016/S0140-6736(20)30154-9. Epub 2020 Jan 24. PMID 31986261
- [Result] Al-Sarraf N, Thalib L, Hughes A, Tolan M, Young V, McGovern E. Effect of smoking on short-term outcome of patients undergoing coronary artery bypass surgery. Ann Thorac Surg. 2008 Aug;86(2):517-23. doi: 10.1016/j.athoracsur.2008.03.070. PMID 18640326
- [Result] Grabas MP, Hansen SM, Torp-Pedersen C, Boggild H, Ullits LR, Deding U, Nielsen BJ, Jensen PF, Overgaard C. Alcohol consumption and mortality in patients undergoing coronary artery bypass graft (CABG)-a register-based cohort study. BMC Cardiovasc Disord. 2016 Nov 11;16(1):219. doi: 10.1186/s12872-016-0403-3. PMID 27835965
- [Result] Guo P. Preoperative education interventions to reduce anxiety and improve recovery among cardiac surgery patients: a review of randomised controlled trials. J Clin Nurs. 2015 Jan;24(1-2):34-46. doi: 10.1111/jocn.12618. Epub 2014 Jun 3. PMID 24894181
- [Result] Hulzebos EH, Helders PJ, Favie NJ, De Bie RA, Brutel de la Riviere A, Van Meeteren NL. Preoperative intensive inspiratory muscle training to prevent postoperative pulmonary complications in high-risk patients undergoing CABG surgery: a randomized clinical trial. JAMA. 2006 Oct 18;296(15):1851-7. doi: 10.1001/jama.296.15.1851. PMID 17047215
- [Result] Mariscalco G, Wozniak MJ, Dawson AG, Serraino GF, Porter R, Nath M, Klersy C, Kumar T, Murphy GJ. Body Mass Index and Mortality Among Adults Undergoing Cardiac Surgery: A Nationwide Study With a Systematic Review and Meta-Analysis. Circulation. 2017 Feb 28;135(9):850-863. doi: 10.1161/CIRCULATIONAHA.116.022840. Epub 2016 Dec 28. PMID 28034901
- [Result] Navaratnarajah M, Rea R, Evans R, Gibson F, Antoniades C, Keiralla A, Demosthenous M, Kassimis G, Krasopoulos G. Effect of glycaemic control on complications following cardiac surgery: literature review. J Cardiothorac Surg. 2018 Jan 17;13(1):10. doi: 10.1186/s13019-018-0700-2. PMID 29343294
- [Result] Marmelo F, Rocha V, Moreira-Goncalves D. The impact of prehabilitation on post-surgical complications in patients undergoing non-urgent cardiovascular surgical intervention: Systematic review and meta-analysis. Eur J Prev Cardiol. 2018 Mar;25(4):404-417. doi: 10.1177/2047487317752373. Epub 2018 Jan 17. PMID 29338307
- [Derived] Scheenstra B, van Susante L, Bongers BC, Lenssen T, Knols H, van Kuijk S, Nieman M, Maessen J, Van't Hof A, Sardari Nia P; DCC Trial Investigators. The Effect of Teleprehabilitation on Adverse Events After Elective Cardiac Surgery: A Randomized Controlled Trial. J Am Coll Cardiol. 2025 Mar 4;85(8):788-800. doi: 10.1016/j.jacc.2024.10.064. Epub 2024 Oct 11. PMID 39396714
- See also: Neil M Ferguson et al. Impact of non-pharmaceutical interventions (NPIs) to reduce COVID-19 mortality and healthcare demand. — https://www.imperial.ac.uk/media/imperial-college/medicine/sph/ide/gida-fellowships/Imperial-College-COVID19-NPI-modelling-16-03-2020.pdf